CLINICAL TRIAL: NCT03558971
Title: Patient Self-administration of Cortisol for Cortisol-responding Disorders in Men and Women Over the Age of 17, Demonstration of Double-blind Trial Results
Brief Title: Patient Self-administration of Cortisol for Cortisol-responding Disorders in Men and Women Over the Age of 17
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Helen Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HF 101
Record Dates: First submitted 2018-05-03; First posted 2018-06-15 (Actual); Last update posted 2018-06-15 (Actual); Status verified 2018-05

CONDITIONS: Rheumatic Diseases
Keywords: Cortisol
MeSH Terms: conditions — Rheumatic Diseases | interventions — Hydrocortisone

STUDY DESIGN:
Intervention Model Description: All participants follow the same treatment protocol: First, the participants ingest a defined dosage, 3-week treatment of cortisol tablets to achieve a minimum symptom state. Second, after the first is complete, participants are trained to self-administer small-dosage, 5-day regimens of cortisol tablets to quench disease exacerbations to maintain the minimum symptom state.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patient self-administration of cortisol (Experimental): Intervention is patient self-administration of cortisol.
  Interventions: Drug: Cortisol

INTERVENTIONS:
Drug: Cortisol — Participants determine when to administer 5-day regimens of cortisol
  Other Names: microdose therapy

SUMMARY:
Participants diagnosed as having fibromyalgia, osteoarthritis, and rheumatoid arthritis are to be brought to a minimum symptom state using a 3-week period during which they are to ingest modest doses of cortisol tablets with weekly lowered tapered doses. Thereafter, the participants are to be taught to self-administer cortisol tablets on the as-needed basis to maintain the minimum symptom state. For this, they are to ingest a smaller-dosage, 5-day tapered regimen of cortisol tablets to quench each reoccurring exacerbation of the disease at its earliest stage. Participants are limited to using less than the safe use limit of cortisol per month and are required to include a minimum of 10 days per month during which no cortisol was ingested.

DETAILED DESCRIPTION:
OBJECTIVE: To define why and demonstrate how patient self-administration of cortisol with stress management eliminates chronic inflammation pain within fibromyalgia, osteoarthritis, and rheumatoid arthritis.

METHODS: One thousand seventeen hundred and twenty (1,720) participants with chronic inflammation-containing diseases, were brought to a minimum symptom state using daily-administered cortisol tablets. Thereafter, participants used 5-day, small-dosage cortisol regimens to quench subsequent disorder exacerbations to maintain the minimum symptom state. Stressors as emotional traumas, infections, allergies, and injuries were minimized to reduce cortisol consumption and participant discomfort. This protocol is compliant with current United States Food and Drug Administration recommendations for cortisol use applied to corticosteroid-responding disorders.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnoses of fibromyalgia, osteoarthritis, or rheumatoid arthritis -

Exclusion Criteria:

Congestive heart failure, stomach ulceration, unstable diabetes, and bipolar disorder

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2430 (Actual)
Dates: Start 2000-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Participant evaluation of disease symptom intensity | Participants determine Total Scores 7 days prior to cortisol initiation to obtain the average baseline Total Score. Participant Total Score change is plotted daily vs. time for study. Outcome: Total Score at 24 weeks vs. baseline.
  Participants evaluate 50 symptoms for intensity using the 0 to 10 scale. 0 represents no disease intensity and 10 represents extreme maximum symptom intensity with the intermediate numbers defined as Mild I, Mild II, Mild III, Moderate I, Moderate II, Moderate III, Severe I, Severe II, Severe III for 2 through 9, respectively. The participant-determined disease intensity numbers of the 50 symptoms are added to obtain Total Score for each day.

CONTACTS AND LOCATIONS:
Overall Officials: Virgil I Stenberg, Ph.D., Principal Investigator — University of North Dakota
Locations (1):
- Helen Foundation Clinic, Apache Junction, Arizona, United States

IPD SHARING:
Plan to Share IPD: No
Plan to publish the study, its results and conclusions

REFERENCES:
- [Background] Stenberg VI, Fiechtner JJ, Rice JR, Miller DR, Johnson LK. Endocrine control of inflammation: rheumatoid arthritis double-blind, crossover clinical trial. Int J Clin Pharmacol Res. 1992;12(1):11-8. PMID 1526694
- [Derived] Irwin JB, Baldwin AL, Stenberg VI. General theory of inflammation: patient self-administration of hydrocortisone safely achieves superior control of hydrocortisone-responding disorders by matching dosage with symptom intensity. J Inflamm Res. 2019 Jun 13;12:161-166. doi: 10.2147/JIR.S195165. eCollection 2019. PMID 31354330